CLINICAL TRIAL: NCT01327235
Title: A Randomized Controlled Multicenter Trial of Endostar and/or Cisplatin in Patients With Malignant Pleural Effusion or Ascites
Brief Title: Endostar and/or Cisplatin for Treatment of Malignant Pleural Effusion or Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-90
Record Dates: First submitted 2011-03-28; First posted 2011-04-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Malignant Pleural Effusion; Malignant Ascites
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — endostar protein; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endostar (Active Comparator)
  Interventions: Drug: Endostar
- Cisplatin (Active Comparator)
  Interventions: Drug: Cisplatin
- Endostar and Cisplatin (Experimental)
  Interventions: Drug: Endostar; Drug: Cisplatin

INTERVENTIONS:
Drug: Endostar — intrapleural injection 45 mg; intraperitoneal injection 60 mg, q3d ×3(d1、d4、d7), 3 times as one cycle, at most 2 cycles
  Arms: Endostar; Endostar and Cisplatin
Drug: Cisplatin — cisplatin 40 mg, q3d ×3(d1、d4、d7), 3 times as one cycle, at most 2 cycles
  Arms: Cisplatin; Endostar and Cisplatin

SUMMARY:
The objective of this study is to compare the efficacy of Endostar/cisplatin with cisplatin alone or Endostar alone in patients with malignant pleural effusion or ascites.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of thoracic or abdominal tumor
* At least medium amount of malignant pleural effusion or ascites
* ECOG Performance Status 0-2
* Life expectancy ≥ 2 months
* Adequate hematologic, cardiac, renal, and hepatic function
* No major surgery within 4 weeks prior to this study
* Written informed consent

Exclusion Criteria:

* Patients with central nervous system (CNS) metastases
* Evidence of bleeding diathesis, serious infection
* Evidence of myocardial infarction, unstable angina or cardiac insufficiency
* Presence of serious COPD and/or respiratory failure
* Allergic to study drug
* Pregnant or lactating women
* Participation in other clinical trials within 30 days prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | baseline to measured progressive disease, every three weeks
  WHO criteria

SECONDARY OUTCOMES:
Time to Progression | baseline to every three weeks until disease progression
Quality of Life | baseline to every three weeks
Incidence of Adverse Events | Up to 1 month after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, MD, Principal Investigator — The 81st Hospital of Chinese PLA
Locations (3):
- China (3):
  - The 81st Hospital of Chinese PLA, Nanjing
  - The Affiliated Hospital of Medical College, QingDao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai